CLINICAL TRIAL: NCT04541823
Title: A Study Evaluating the Effect of Desflurane in Preventing Postoperative Cognitive Dysfunction
Brief Title: The Effect of Desflurane on Postopertative Cognitive Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Anshi Wu, Head of Anesthesiology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00375928
Record Dates: First submitted 2020-08-04; First posted 2020-09-09 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane (Experimental): Patients allocated to this arm will receive desflurane during the maintenance of anesthesia.
  Interventions: Drug: Desﬂurane
- Propofol (Placebo Comparator): Patients allocated to this arm will receive propofol during the maintenance of anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desﬂurane — Investigators administrated desflurane with target of BIS 40-60 during the maintenance of anesthesia
  Arms: Desflurane
Drug: Propofol — Investigators administrated propofol with target of BIS 40-60 during the maintenance of anesthesia
  Arms: Propofol

SUMMARY:
The purpose of this study is to determine the effect of desflurane on postoperative cognitive dysfunction

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction is a common complication during postoperative period，especially in elderly patients. It is characterized by cognitive decline, inattention and abnormal mental status following surgery. The presence of postoperative cognitive dysfunction is independently associated with poor recovery, increased hospital length of stay and increased mortality.

Desflurane is a widely used volatile anesthetic, associated with shorter emergence times than other volatile anesthetics. This study aims to access the effect of desflurane in preventing postoperative cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written consent given
* 2. Scheduled to undergo elective non-cardiac surgeries under general anesthesia
* 3. ASA Physical Score I-III

Exclusion Criteria:

* 1. Patients with a history of neurological disease, such as Alzheimer disease.
* 2. Patients with a history of psychiatric disease
* 3. Patients with a medication history of antipsychotic drugs.
* 4. Unable to complete neuropsychological testing including patients with severe visual or hearing impairment.
* 5. Patients with preoperative delirium.
* 6. Patients who have severe adverse events, such as cardiac arrest.
* 7. Patients who preoperative MMSE score are below 20;
* 8. Patients who undergo second operation in a short period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction | on the 30th day after surgery
  Screening of the patients regarding an postoperative cognitive dysfunction by TICS-M.TICS-M is assessed at 30 days after surgery

SECONDARY OUTCOMES:
Incidence of postoperative delirium | 1-7days after surgery, on the 30th day after surgery
  Screening of the patients regarding a postoperative delirium by The Confusion Assessment Method for The Intensive Care Unit (CAM-ICU)
Postoperative Pain | Within 3 days after surgery
  Visual Analogue Scale will be used to assess postoperative pain of patients. Numerical rating scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain.
EEG frequency spectrum | 5 minutes before anesthesia introduction to 5 minutes before discharge from PACU
  Electroencephalography will be recorded at different points of time as follows and EEG characteristics including power in alpha, beta, theta, delta, gamma, spectrum will be extracted using MATLAB:
  1. Five minutes before anesthesia introduction
  2. During the entire operation
  3. At discharge from post-anesthesia care unit (PACU)
Mortality | Within 30 days after surgery
Length of Hospital stay | From the date of admission until discharged from hospital, within 30 days
Hospital readmission | Within 30 days after surgery
  Hospital readmission during the follow up
Incidence of postoperative nausea and vomiting | Within 7 days after surgery
Adverse events | Within 30 days after surgery
  Other adverse events within 3 days after surgery were noted
Neural and hemodynamic responses during desflurane general anesthesia | 5 minutes before anesthesia introduction to 5 minutes after emergence
  Functional near-infrared spectroscopy (fNIRS) will be monitored from pre-anesthesia to the emergence. △[HbO] ，△[Hb] will be recorded. Besides, the coupling of fNIRS signals with neuronal signals (EEG) will be calculated. Furthermore, sample entrophy and the phase difference between △[HbO] and △[Hb] will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China